CLINICAL TRIAL: NCT00821587
Title: Cyclosporine in Hepatitis C Infection Viral Clearance Following Liver Transplantation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20040658
Record Dates: First submitted 2009-01-09; First posted 2009-01-13 (Estimated); Results first posted 2011-12-08 (Estimated); Last update posted 2023-06-01 (Actual); Status verified 2023-05

CONDITIONS: Hepatitis C
Keywords: Hepatitis C Post Liver Transplant
MeSH Terms: conditions — Hepatitis C | interventions — Cyclosporine; Cyclosporins; Tacrolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tacrolimus (Active Comparator): Tacrolimus
  Interventions: Drug: Tacrolimus
- Cyclosporine (Active Comparator): Cyclosporine
  Interventions: Drug: Cyclosporine

INTERVENTIONS:
Drug: Cyclosporine — Patients randomized to CsA had TAC discontinued and were treated with CsA at a dose of 2.0-4.0 mg/kg/day orally in two divided doses with target trough whole blood concentrations of 150-200 ng/ml.
  Other Names: Gengraf
  Arms: Cyclosporine
Drug: Tacrolimus — Patients receiving TAC were treated with a dose of 0.08-0.12 mg/kg/day orally in two divided doses with target trough whole blood concentrations of 10-15 ng/ml for the first month post-transplant followed by 5-10 ng/ml thereafter. Immunosuppression was typically tapered to monotherapy (TAC alone) within 4-6 months of transplantation.
  Other Names: Prograf
  Arms: Tacrolimus

SUMMARY:
The purpose of this study is to evaluate the effect of cyclosporine, an anti-rejection drug, on the clearance of the hepatitis C virus in liver transplant subjects being treated with peg-interferon and ribavirin.

DETAILED DESCRIPTION:
This is a randomized, single-center controlled study comparing two different immunosuppression regimens (CsA and TAC) in patients with recurrent HCV after LT undergoing antiviral therapy for HCV.

ELIGIBILITY:
Inclusion Criteria:

* Males and females age 18 years and older
* HCV RNA positive by PCR after liver transplantation
* Elevated ALT at any time point after liver transplantation
* Protocol liver biopsy (standard of care) consistent with Stage greater than or equal to 2 of Ishak fibrosis score after liver transplantation
* Able to provide written informed consent
* Willing to practice acceptable birth control during the study period.

Exclusion Criteria:

* Decompensated Cirrhosis
* hemoglobin < 12 g/dl
* WBC < 3,500/cubic mm
* Platelets < 75,000/cubic mm
* Human immunodeficiency virus infection
* Pregnancy
* Positive HbsAg
* History of coronary artery disease, history of seizure disorder, poorly controlled autoimmune conditions, thyroid dysfunction, diabetes mellitus, major psychosis, intolerance to previous interferon-based therapy other than anemia or neutropenia
* History of suicidal ideation or suicidal attempts
* Creatinine > 2.0 mg/dl
* Severe non-hepatic illnesses

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2004-06; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Roberto J Firpi-Morell, MD, Principal Investigator — University of Florida

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at the University of Florida in Gainesville between July 2004 and April 2008. Patients attended clinic visits at the time of randomization (baseline) and at 12-week intervals for 72 weeks.
Pre-assignment Details: Subjects with Hepatitis C Virus (HCV) recurrence Ishak Stage2 were enrolled and randomized to stay on Tacrolimus (TAC) or to change to Cyclosporine (CsA) for baseline immunosuppression with 1-month washout period before initiation of therapy with Pegylated Interferon Alfa2a and ribavirin for 48 weeks for genotype-1, or 24 weeks for genotype-3.
Groups:
- Tacrolimus: Patients receiving TAC are treated with a dose of 0.08- 0.12 mg/kg/day orally in two divided doses with target trough whole blood concentrations of 10-15 ng/ml for the first month post-transplant followed by 5-10 ng/ml thereafter.
- Cyclosporine: Patients randomized to CsA will have TAC discontinued and will be treated with CsA at a dose of 2.0-4.0 mg/kg/day orally in two divided doses with target trough whole blood concentrations of 150-200 ng/ml.
Period: Overall Study
Arm/Group | Tacrolimus | Cyclosporine
Started | 20 | 19
Completed | 20 | 18
Not Completed | 0 | 1
Not completed — Physician Decision | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Tacrolimus | Cyclosporine | Total
Number analyzed (Participants) | 20 | 19 | 39
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 20 | 19 | 39
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.4 (5.4) | 52.2 (6.4) | 53.3 (5.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 5 | 7
  Male | 18 | 14 | 32
Region of Enrollment [Number; unit: participants]
  United States | 20 | 19 | 39

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Less Than 100 Hepatitis C Virus RNA Copies/mL
Description: Number of Participants with Undetectable or Less than 100 copies/ml Hepatitis C Viral Level --defined as SVR -Sustained Virologic Response
Time Frame: 6 months after completion of interferon based therapy
Population: Randomization was performed using computer-generated random numbers. 150 patients were eligible and 39 met entry criteria for enrollment in the study. Subjects with HCV recurrence (Ishak Stage2) were randomized to TAC or to change to CsA before initiation of therapy with PEGa-2a and ribavirin for 48 weeks for genotype-1,or 24 weeks for genotype-3.
Measure: Count of Participants; unit: Participants
Groups:
- Tacrolimus (TAC): Tacrolimus 0.08-0.12 mg/kg/day orally in two divided doses
- Cyclosporine (CsA): Cyclosporine 2.0-4.0 mg/kg/day orally in two divided doses
Arm/Group | Tacrolimus (TAC) | Cyclosporine (CsA)
Number analyzed (Participants) | 20 | 18
Participants | 7 | 7
Statistical Analysis 1: Comparison: Tacrolimus (TAC) vs Cyclosporine (CsA); We hypothesize that subjects on CsA are more likely to achieve undetectable viral levels after liver transplant. Comparisons between the two groups (Undetectable viral level vs. Detectable viral level) were performed with Pearson Chi-square tests or Fisher's exact test for categorical variables, and Mann-Whitney U test for continuous variables; Test type: Superiority or Other; p < 0.05, Chi-squared — We hypothesize that subjects on CsA are more likely to achieve undetectable viral level in patients receiving antiviral therapy for recurrent HCV after Liver Transplant

ADVERSE EVENTS:
Time Frame: 72 weeks
Arm/Group | Tacrolimus | Cyclosporine
Serious Adverse Events (participants affected / at risk) | 0/20 | 1/19
Other Adverse Events (participants affected / at risk) | 16/20 | 17/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tacrolimus (N=20) | Cyclosporine (N=19)
Death (Immune system disorders) | 0 (0) | 1 (1) — Liver biopsy was performed and showed severe chronic rejection
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tacrolimus (N=20) | Cyclosporine (N=19)
Neutropenia (Blood and lymphatic system disorders) | 8 (8) | 3 (4) — Labs
Anemia (Blood and lymphatic system disorders) | 16 (20) | 16 (19) — Labs
Thrombocytopenia (Blood and lymphatic system disorders) | 11 (11) | 10 (10) — Labs
Depression (Psychiatric disorders) | 8 (8) | 9 (9) — Clinical Assessment
Nausea (Gastrointestinal disorders) | 5 (8) | 5 (10) — Reported by patient
Fever (General disorders) | 4 (16) | 4 (20) — Reported by patient
Insomnia (General disorders) | 6 (6) | 9 (9) — Reported by patient
Irritability (Psychiatric disorders) | 2 (6) | 3 (5) — Reported by patient

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No